CLINICAL TRIAL: NCT03262792
Title: A Double-blind, Randomized, Placebo Controlled Study to Assess the Efficacy of Andrographis Paniculata in Subjects With Mild to Moderate Osteoarthritis Over a 12-weeks Period
Brief Title: Assessment of the Efficacy of Andrographis Paniculata in Subjects With Mild to Moderate Osteoarthritis
Acronym: A Paniculata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VL/170105/PA/OA
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Andrographis paniculata extract

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled, parallel groups study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo
- Andrographis Paniculata 150 (Active Comparator): Andrographis Paniculata 150 mg
  Interventions: Dietary Supplement: Andrographis Paniculata
- Andrographis Paniculata 300 (Active Comparator): Andrographis Paniculata 300 mg
  Interventions: Dietary Supplement: Andrographis Paniculata

INTERVENTIONS:
Dietary Supplement: Placebo — Microcrystalline cellulose
  Arms: Placebo
Dietary Supplement: Andrographis Paniculata — Andrographis Paniculata 150 mg
  Arms: Andrographis Paniculata 150
Dietary Supplement: Andrographis Paniculata — Andrographis Paniculata 300 mg
  Arms: Andrographis Paniculata 300

SUMMARY:
This is a 12 weeks randomized, double-blind, placebo-controlled clinical study to assess the effect of Andrographis Paniculata at low dose of 300 mg/day and high dose of 600 mg/day in the study population in the age range of 40-70 years and suffering from mild-moderate OA.

DETAILED DESCRIPTION:
In this study, we will assess the efficacy parameters such as effect on various joint health parameters (pain, stiffness and physical activity) by using WOMAC scale. The individuals with knee OA suffer from an increased impact on their activities of daily living, which leads to losses in labor relations, leisure, social life, and sleeping quality, leading also to important decrease in their quality of life. Thus, an important outcome to be evaluated in this study is quality of life of these individuals which will be assessed by SF-36 self-reported questionnaire. One of the aims of this study is therefore to investigate the levels of different dimensions of fatigue in knee OA and to assess changes in fatigue after the treatment targeting pain reduction and physical functioning by the use of FACIT-fatigue questionnaire.

Effect of the treatment on rescue medication consumption which is directly proportional to the degree of pain will also be captured via this study. The hepatic (SGOT and SGPT) and renal (serum creatinine) safety biomarkers will be assessed to investigate the effect of chronic use of Andrographis Paniculata on liver and kidneys.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects in the age range of 40 - 70 years (both inclusive).
2. Body mass index (BMI) must be ≥ 25 and < 29.9 kg/m2.
3. Radiographic evidence of grade I- II osteoarthritis of knee joint, based on the Kellgren and Lawrence radiographic entry criteria with WOMAC pain score in range of 10-16.
4. History of primary idiopathic osteoarthritis of the knee characterized by pain of mild to moderate intensity which requires intake of analgesics.
5. Self-reported difficulty in at least one of the following activities attributed to knee pain: walking a distance of 400 metres, getting in and out of the car, going up and down the stairs or stiffness observed in the knee if > 30 minutes in the same position.
6. Female subjects of child-bearing age must be willing to use the accepted methods of contraception during the course of the study.
7. Ability to provide written informed consent.

Exclusion Criteria:

1. Prior or ongoing medical conditions (e.g. concomitant illness, psychiatric condition, alcoholism, drug abuse), medical history, physical findings, ECG findings or laboratory abnormalities that in the investigator's opinion could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed or could impair the assessment of study results.
2. History of surgery or major trauma to the study joint.
3. History of arthroscopic surgery or intervention on the study joint.
4. Subjects who have received intra-articular steroids or hyaluronic acid within the last three months.
5. Signs of active study joint inflammation including redness, warmth, and/or, if qualifying with osteoarthritis of the knee, a large, bulging effusion of the study knee joint with the loss of normal contour of the joint at the screening visit or at the baseline examination after the washout period.
6. Subjects awaiting a replacement of knee or hip joint.
7. Subjects with other conditions that cause pain.
8. Subjects with deformity of the knee joint.
9. Subject who are significantly incapacitated or disabled and would be categorized as ACR Functional Class IV (largely or wholly incapacitated), or unable to walk without assistive devices.
10. Subjects with other known rheumatic or inflammatory disease such as rheumatoid arthritis, osteomyelitis and bone metastasis.
11. Other pathologic lesions on X-rays of knee.
12. Positive hepatitis B surface antigen, Hepatitis C antibody, Anti human immunodeficiency virus (HIV) antibody test, or VDRL.
13. History of bleeding disorders.
14. Inability to comply with the protocol requirements.
15. Participation in any other clinical trial within 3 months of registering in this trial.
16. Women of child-bearing potential with a positive pregnancy test or who are lactating.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
WOMAC pain score | 84 days
  Change in WOMAC pain score

SECONDARY OUTCOMES:
WOMAC stiffness score | 84 days
  Change in WOMAC stiffness score
WOMAC physical function score | 84 days
  Change in WOMAC physical function score
SF-36 | 84 days
  Change in SF-36's various component scores.
FACIT score | 84 days
  Change in FACIT score
Rescue medication consumption | 84 days
  Change in rescue medication consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Srivastava, MD, Study Director — Vedic Lifesciences
Locations (4):
- India (4):
  - Nidaan Hospital, A/1, Adinath Society, Near Dosti Estate, Opposite Antop Hill Post Office, Wadala(West), Mumbai, Maharashtra
  - Ayush nursing Home, Gaurav vista, Gaurav Garden,BunderpakhadiRoad, Kandivali(West), Mumbai, Maharashtra
  - Siddhant Clinic, Shop No. 17, Lenyadri Cooperative Housing Society, Sector 19A, Nerul(East),Navi Mumbai -400706, Maharashtra, Mumbai, Maharashtra
  - Orthopaedic Clinic, 213, 2nd floor, Shiv Centre, Plot no. 72, Sector-17, Vashi, Navi Mumbai., Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://hpingredients.com/products/premier-ingredients/paractin/